CLINICAL TRIAL: NCT02223130
Title: Addressing Discrimination and Mistrust Among Black Men: Phase III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Fenway Community Health (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura Bogart, Associate Professor of Pediatrics, Harvard Medical School; Research Director, Division of General Pediatrics, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00002878; R34MH096544-03 (NIH)
Record Dates: First submitted 2014-08-12; First posted 2014-08-22 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: HIV
Keywords: HIV; Discrimination; Coping; Medical Mistrust; HIV Outcomes; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Participants will attend the baseline, first follow-up, and final follow-up study visits, at which they take computer surveys. After their baseline interview and before their first follow-up interview, participants attend the Intervention Group, which consist of 9 weekly group sessions. Each of the weekly sessions is led by a mental health professional and a peer facilitator who uses Cognitive Behavioral Therapy techniques to work with participants in tracking their cognitions, emotions, and behaviors in response to stressful/discrimination experiences.
  Interventions: Behavioral: Cognitive Behavioral Therapy techniques
- Waitlist Control (No Intervention): Participants are not given the Intervention Group while they are enrolled in the study. Instead, they only attend the baseline, first follow-up, and final follow-up study visits, at which they take computer surveys.
  After they have completed the study, participants from the first two cohorts are offered the option of attending an intervention group that is identical in content to the intervention group being studied.The third cohort is offered the intervention group after they have completed the first follow-up but before they complete the final follow-up due to timing and budgetary restraints. No data is collected and no incentives are given during these intervention groups.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy techniques — Participants attend 9 weekly group sessions. Each of the weekly sessions is led by a mental health professional and a peer facilitator who use Cognitive Behavioral Therapy techniques to work with participants in tracking their cognitions, emotions and behaviors in response to stressful/discrimination experiences.
  Arms: Intervention Group

SUMMARY:
The purpose of this research study is to test a group program aimed at improving the quality of life of HIV+ Black men who have sex with men. The group will address ways to cope with discrimination and will help men examine mistrust that they may have about healthcare, including doctors and other healthcare providers and HIV medications. The aim is to provide a supportive community for HIV+ Black men.

DETAILED DESCRIPTION:
The aim of the study is to examine whether the pilot intervention can reduce mistrust and improve coping responses to discrimination among HIV positive Black men who have sex with men (MSM). We will conduct a small randomized pilot trial to test the feasibility of evaluation methods. All participants will attend a baseline, a first follow-up visit, and a final follow-up visit (each 3 months apart) at which they will take computer assessments. Participants who are assigned to the intervention will attend 9 weekly intervention sessions after baseline and before the first follow-up. Using a wait-list control design, control group participants from the first two cohorts will be offered the intervention after they complete the final follow-up visit. Control group participants from the third cohort will be offered the intervention after they complete the first final-up visit and before they complete their final follow-up due to timing and budgetary restraints. We will hold three consecutive groups for our small randomized control trial. This means that we will be recruiting continuously; once we finish recruiting for the first group, we will start recruiting for the second group, and so on. Each group has about 12 or 13 intervention and 7-11 control participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older
* Biologically male at birth
* Currently self-identifies as male
* Self-identifies as Black or African American (mixed-race individuals will be eligible if they primarily identify as Black or African American)
* HIV-positive
* Reported having sex with men in lifetime
* Able and willing to provide informed consent

Exclusion Criteria:

* Does not meet all of the inclusion criteria (e.g., if they are unable to provide proof of their HIV-positive status)
* Unable to provide informed consent
* Reports or presents evidence of severe mental health problems that require immediate treatment (e.g., psychotic symptoms, active suicidality at time of enrollment) or diagnosed mental disorder that would limit the ability to participate (e.g., dementia)
* Reports or presents evidence of cognitive impairments that limit the ability to comprehend the informed consent or to fully participate in the various parts of the study (assessments, intervention, homework).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Coping | 3 months post-baseline
  Improved coping scores on Brief Cope, Emotional and Behavioral Coping, and Africultural Coping scales

SECONDARY OUTCOMES:
Mistrust | 3 months post-baseline
  Reduced mistrust scores on Medical Mistrust scale

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Bogart, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Fenway Health, Boston, Massachusetts, United States